CLINICAL TRIAL: NCT06778031
Title: An Open, Multicenter Phase II Clinical Study of SHR-A1811 in the Treatment of HER2-positive Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: A Clinical Study of SHR-A1811 in the Treatment of HER2-positive Locally Advanced or Metastatic Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-215
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Locally Advanced or Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The SHR-A1811 combination group (Experimental)
  Interventions: Drug: SHR-A1811; Drug: SHR-1316; Drug: SHR-8068

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811.
Drug: SHR-1316 — SHR-1316.
Drug: SHR-8068 — SHR-8068.

SUMMARY:
This study is an open, multicenter Phase II clinical trial to evaluate the efficacy and safety of the SHR-A1811 combination in HER2 positive patients with locally advanced or metastatic biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including both ends), male or female;
2. ECOG-PS score: 0 or 1;
3. Expected survival ≥ 12 weeks;
4. Locally advanced or metastatic biliary tract cancer confirmed by histopathology or cytology;
5. Subjects who had not previously received any systemic antitumor therapy were allowed to have previously received radical therapy, and had received the last dose of radical therapy for at least 6 months until disease recurrence;
6. According to the RECIST v1.1 standard, the subjects had at least one measurable lesion;
7. The main organ function is normal, in line with the program requirements;
8. Consent to contraception.

Exclusion Criteria:

1. Other active malignancies within 5 years or at the same time;
2. Local antitumor therapy was received within 4 weeks prior to initiation of treatment;
3. Subjects with biliary obstruction should be excluded;
4. There is active autoimmune disease or a history of autoimmune disease that may recur;
5. Known or suspected history of interstitial pneumonia or interstitial lung disease, or prior history of interstitial pneumonia or interstitial lung disease requiring hormone therapy;
6. Severe infection within 4 weeks prior to initiation of study treatment;
7. Active hepatitis B virus (HBV) infection;
8. Have serious cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of the SHR-A1811 combination evaluated by investigators | Screening up to study completion, an average of 3 year.

SECONDARY OUTCOMES:
Duration of response (DoR) of the SHR-A1811 combination evaluated by investigators | Screening up to study completion, an average of 3 year.
Disease control rate (DCR) of the SHR-A1811 combination evaluated by investigators | Screening up to study completion, an average of 3 year.
Progression free survival (PFS) of the SHR-A1811 combination evaluated by investigators | Screening up to study completion, an average of 3 year.
Overall survival (OS) of the SHR-A1811 combination evaluated by investigators | Screening up to study completion, an average of 3 year.
Adverse events (AEs) | Screening up to study completion, an average of 3 year.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided